CLINICAL TRIAL: NCT01554501
Title: The Role of Stress in Self-Control, Coping and Emotion Regulation
Brief Title: The Role of Stress in Self-Control, Coping, and Emotion Regulation
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rajita Sinha, Professor, Yale University
Other Study IDs: 0710003159; 5PL1DA024859-05 (NIH)
Record Dates: First submitted 2012-03-01; First posted 2012-03-15 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Stress
Keywords: stress; self-control; emotion regulation; health
MeSH Terms: conditions — Self-Control; Emotional Regulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood taken for understanding genetic factors.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Community sample

SUMMARY:
The purpose of this study is to examine the effects of stress on mental and physical health and behavior.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-50
* able to read and write

Exclusion Criteria:

* Any psychotic disorder or current psychiatric symptoms requiring specific attention, including active symptoms of psychosis or suicidal/homicidal ideation
* Pregnant women
* Inability to give informed consent
* Traumatic brain injury or loss of consciousness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 855 (Actual)
Dates: Start 2007-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Stress response and lifestyle behaviors | Baseline
  Study explores differences in measures of stress as they relate to self-control, coping, emotion regulation and lifestyle and health outcomes.

SECONDARY OUTCOMES:
Biological stress responses | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Stress Center, New Haven, Connecticut, United States